CLINICAL TRIAL: NCT02135757
Title: A Phase IV Multicenter Trial to Evaluate Real-world Health Outcomes, Economic Impact and Resistance Mechanisms of Panitumumab in the Treatment of Patients With Chemotherapy-refractory Metastatic Colorectal Cancer
Brief Title: Study to Evaluate Real-world Pharmacoeconomics and Resistance Mechanisms of Panitumumab in Metastatic Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: PeriPharm (Other)
Collaborators: Personalized Medicine Partnership for Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: PMPC-02
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a phase IV multicenter trial to evaluate real-world health outcomes, economic impact and resistance mechanisms of panitumumab in the treatment of patients with chemotherapy-refractory metastatic colorectal cancer (mCRC).

This study will address two anticipated issues surrounding personalized medicine and treatment with panitumumab. First, it will enable to assess the economic impact of panitumumab in a real-life setting (HEOR study). Second, it will identify new blood-based mechanisms of resistance, which may lead to new avenues for combination therapy in metastatic colorectal cancer (Blood study).

The primary objective is to collect information on quality of life and health care resource utilization by patients diagnosed with metastatic colorectal cancer. The secondary objectives are to confirm survival data, to assess the quality of life of patients and to assess the health care resource utilization of patients. The blood biomarker study objective is to determine blood-based biomarkers of response or resistance to panitumumab.

Patients with a mutated KRAS gene will be treated with standard-of-care (SOC) and will participate to the HEOR study only. Patients with a non-mutated (wild type) KRAS gene will be treated with panitumumab and will participate to the HEOR study and to the blood biomarker study.

During the course of the study, data will be collected on quality of life and work productivity. Patients will be asked to fill a set of questionnaires at their recruitment in the study and at every 3 months after treatment initiation. For patients participating to the blood study (patients with a wild type KRAS), blood samples will be collected before patients start their treatment, at every treatment and when they discontinue their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of mCRC.
* Immunohistochemical evidence of EGFR expression.
* ECOG performance status of 0, 1 or 2.
* Patients refractory to fluoropyrimidine, oxaliplatin, and irinotecan chemotherapy regimens
* Patients with a wt KRAS scheduled to receive panitumumab as a single agent for the third-line treatment of mCRC or patients with a mt KRAS scheduled to receive SOC for third-line treatment of mCRC.
* Signed and dated IRB-approved informed consent document.
* Ability to read and understand English or French.
* 18 years of age or older.

Exclusion Criteria:

* Acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chemotherapy-refractory metastatic colorectal cancer from participating hospitals in Quebec.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-08; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The pharmacoeconomic impact of panitumumab for the treatment of metastatic colorectal cancer in a real-life setting | From the date of registration until date of death from any cause, assessed up to 38 months.
  Pharmacoeconomic impact (cost-effectiveness and cost-utility) will be evaluated by questionnaires completed by the patient and caregiver. These include quality of life, health resource utilization, work productivity and activity impairment, and health questionnaires.

SECONDARY OUTCOMES:
Identification of blood biomarkers that confer significant improvement in progression-free survival in patients treated with panitumumab. | From the date of registration until the date of disease progression, assessed up to 24 months (estimation).
  Plasma will be isolated from patients pre-treatment, at every disease assessment and at progression of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lachaine, PhD, Principal Investigator — PeriPharm
Locations (2):
- Canada (2):
  - Hôpital Charles-Le Moyne, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec